CLINICAL TRIAL: NCT02357732
Title: A Phase I Study of the Anti-PD-1 Antibody Nivolumab in Combination With Dabrafenib and/or Trametinib in Patients With BRAF or NRAS-mutated Metastatic Melanoma
Brief Title: Study of the Anti-PD-1 Antibody Nivolumab in Combination With Dabrafenib and/or Trametinib
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI decided not to proceed
Sponsor: University of Pittsburgh (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Hussein Tawbi, Associate Professor of Medicine, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-115
Record Dates: First submitted 2015-01-27; First posted 2015-02-06 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Metastatic Melanoma
Keywords: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; trametinib; dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nivolumab and Dabrafenib Combination (doublets) (Experimental): Level -1, Nivolumab 1mg/kg IV every 2 weeks (q2 weeks); Dabrafenib 100mg by mouth (PO) twice a day(BID) every day (QD); Level 1, Nivolumab 1mg/kg IV q2 weeks; Dabrafenib 150mg PO BID QD; Level 2, Nivolumab 3mg/kg IV q2 weeks; Dabrafenib 150mg PO BID QD;
  Interventions: Drug: Nivolumab; Drug: Dabrafenib
- Nivolumab and Trametinib Combination (doublets) (Experimental): Level -1, Nivolumab 1mg/kg IV q2 weeks; Trametinib 1mg PO QD; Level 1, Nivolumab 1mg/kg IV q2 weeks; Trametinib 2mg PO QD; Level 2, Nivolumab 3mg/kg IV q2 weeks; Trametinib 2mg PO QD;
  Interventions: Drug: Nivolumab; Drug: Trametinib
- Nivolumab, Dabrafenib and Trametinib Combination (triplet) (Experimental): Level -1, Nivolumab 1mg/kg IV q2 weeks; Dabrafenib 150mg PO BID; Trametinib 1mg PO QD; Level 1, Nivolumab 1mg/kg IV q2 weeks; Dabrafenib 150mg PO BID; Trametinib 2mg PO QD; Level 2, Nivolumab 3mg/kg IV q2 weeks; Dabrafenib 150mg PO BID; Trametinib 2mg PO QD;
  Interventions: Drug: Nivolumab; Drug: Trametinib; Drug: Dabrafenib

INTERVENTIONS:
Drug: Nivolumab
Drug: Trametinib
  Arms: Nivolumab and Trametinib Combination (doublets); Nivolumab, Dabrafenib and Trametinib Combination (triplet)
Drug: Dabrafenib
  Arms: Nivolumab and Dabrafenib Combination (doublets); Nivolumab, Dabrafenib and Trametinib Combination (triplet)

SUMMARY:
This study evaluates nivolumab in combination drug treatments involving 1) nivolumab and dabrafenib 2) nivolumab and trametinib and 3) nivolumab, dabrafenib and trametinib in patients with BRAF or NRAS-mutated metastatic melanoma.

DETAILED DESCRIPTION:
Patients are being asked to take part in this clinical research study because they have BRAF- or NRAS-mutated metastatic melanoma. If they participate they will receive the investigational drug nivolumab in combination with dabrafenib and/or trametinib based on their medical diagnosis, BRAF V600 test results and/or NRAS-mutated status.

The research study will evaluate the safety and efficacy of the two drugs nivolumab and dabrafenib or nivolumab and trametinib. Once this is evaluated, then additional subjects will be enrolled for treatment with the triplicate (all 3 drugs) of nivolumab, dabrafenib and trametinib together.

A treatment cycle will be 28 days, coinciding with the administration of nivolumab. The DLT evaluation period will be restricted to cycle 1, although toxicities in subsequent cycles will be closely evaluated. In trametinib-containing arms, a loading dose will be given on days 1 and 2 of cycle 1 to allow steady state concentrations to be achieved within one week of administration.

In the absence of treatment delays due to adverse event(s), treatment may continue for 3 years or until one of the following criteria applies:

* Disease progression
* Intercurrent illness that prevents further administration of treatment
* Unacceptable adverse event(s)
* Patient decides to withdraw from the study
* General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator

Patients will be considered evaluable for toxicity if they receive 1 complete cycle of therapy, or if they experience dose limiting toxicities (DLTs). Definition of DLTs include:

* Any Grade 2 drug-related uveitis or eye pain or blurred vision that does not respond to topical therapy and does not improve to Grade 1 severity within the re-treatment period OR requires systemic treatment
* Any Grade 3 non-skin, drug-related adverse event lasting > 7 days, with the following exceptions for drug-related laboratory abnormalities, uveitis, pneumonitis, bronchospasm, diarrhea, colitis, neurologic adverse event, hypersensitivity reactions, and infusion reactions
* Grade 3 drug-related uveitis, pneumonitis, bronchospasm, diarrhea, colitis, neurologic adverse event, hypersensitivity reaction, or infusion reaction of any duration requires discontinuation
* Grade 3 drug-related laboratory abnormalities do not require treatment discontinuation except the following: Grade 3 drug-related thrombocytopenia > 7 days or associated with bleeding requires discontinuation; Any drug-related liver function test (LFT) abnormality that meets the following criteria require discontinuation - AST or ALT > 8 x ULN; Total bilirubin > 5 x ULN; Concurrent AST or ALT > 3 x ULN and total bilirubin > 2 x ULN;
* Any Grade 4 drug-related adverse event or laboratory abnormality, except for the following events which do not require discontinuation:

  * Isolated Grade 4 amylase or lipase abnormalities that are not associated with symptoms or clinical manifestations of pancreatitis and decrease to < Grade 4 within 1 week of onset.
  * Isolated Grade 4 electrolyte imbalances/abnormalities that are not associated with clinical sequelae and are corrected with supplementation/appropriate management within 72 hours of their onset
* Any dosing interruption lasting > 6 weeks with the following exceptions:

  * Dosing interruptions to allow for prolonged steroid tapers to manage drug-related adverse events are allowed. Prior to re-initiating treatment in a subject with a dosing interruption lasting > 6 weeks, the Investigator must be consulted. Tumor assessments should continue as per protocol even if dosing is interrupted
  * Dosing interruptions > 6 weeks that occur for non-drug-related reasons may be allowed if approved by the Investigator. Prior to re-initiating treatment in a subject with a dosing interruption lasting > 6 weeks, the Investigator must be consulted. Tumor assessments should continue as per protocol even if dosing is interrupted Any adverse event, laboratory abnormality, or intercurrent illness which, in the judgment of the Investigator, presents a substantial clinical risk to the subject with continued nivolumab dosing.

Patients will be followed for 2 years after removal from study or until death, whichever occurs first, through standard of care visits or by medical records review. Patients removed from study for unacceptable adverse event(s) will be followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic melanoma (Stage IV) or unresectable Stage III melanoma with BRAF V600E/K or NRAS mutations.
* Prior therapies for metastatic melanoma are allowed, including chemo-, cytokine-, immuno-, biological- and vaccine-therapy as long as they did not include BRAFi, MEKi, or nivolumab. Prior ipilimumab therapy will be allowed with a washout period of 8 weeks and if all autoimmune adverse events have resolved to grade 1.
* Evidence of evaluable disease.
* ECOG Performance Status of 0 or 1.
* Stable CNS disease is allowed. Subjects with brain metastases are eligible if (a) metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for 4 weeks after treatment is complete and within 28 days prior to the first dose of nivolumab administration; or (b) if they are untreated but asymptomatic and do not require steroid therapy. Patients are excluded if they require high doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration, as this could result in immunosuppression.
* Patients must have normal organ and marrow function as defined by the normal laboratory ranges. Screening laboratory values must meet the following criteria and should be obtained within 28 days prior to registration:

  * WBC ≥ 2000/μL
  * Neutrophils ≥ 1500/μL
  * Platelets ≥ 100 x103/μL
  * Hemoglobin > 9.0 g/dL
  * Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):

Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL

* AST/ALT ≤ 3 x ULN
* Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)

  * Men and women age≥18 years.
  * Life expectancy of greater than12 weeks.
  * Women of childbearing potential (WOCBP) must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug. WOCBP are those who have not been surgically sterilized or have not been free from menses for > 1 year.
  * Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of nivolumab.
  * Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) and azoospermic men do not require contraception.
  * Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Histologically confirmed metastatic melanoma (Stage IV) with NRAS and BRAF-wild type.
* Grade 3/4 immune-related AEs on ipilimumab and required more than 12 weeks of immune suppression with corticosteroids.
* History of interstitial lung disease or pneumonitis.
* History of known glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Active leptomeningeal metastases or untreated symptomatic brain metastases.
* Active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Require systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Known history of a positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with dabrafenib and trametinib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* History of allergy or adverse drug reaction to the study drug components (nivolumab, dabrafenib, or trametinib) or drugs of similar chemical or biologic composition. Patients with a history of severe hypersensitivity reaction to any monoclonal antibody should also be excluded.
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding women are excluded from this study. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with dabrafenib and trametinib, breastfeeding should be discontinued if the mother is treated with dabrafenib and trametinib. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To determine the Maximally Tolerated Dose and/or Recommended Phase II Dose (RP2D) of nivolumab in combination with dabrafenib and/or trametinib in patients with BRAF- or NRAS-mutated metastatic melanoma | The first four weeks of dosing
  It is planned to determine the maximum tolerable dose with a modified version of the standard "up and down" (3+3) dose-finding method using cohorts of 3 patients. At the start of the trial, three patients will be placed on dose level 1. The decision rules based on the observed dose limiting toxicities (DLTs) in this and subsequent cohorts are given. Only DLTs observed in a patient during the first cycle (28 days) will be used for the dose escalation decisions. Patients will be considered evaluable for toxicity if they receive 1 complete cycle of therapy, or if they experience DLT; in-evaluable patients will be replaced.

SECONDARY OUTCOMES:
Antitumor Effects and Immune Related Response | Every twelve weeks for three years while on study drug
  Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) and by the Immune Related Response Criteria. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Hussein Tawbi, MD, Principal Investigator — University of Pittsburgh Medical Center / Hillman Cancer Center